CLINICAL TRIAL: NCT00577603
Title: A Controlled, Randomized Study to Evaluate and Compare the Rate of Para-Stomal Herniation After Permanent Stoma Formation With and Without Reinforcement With a Collagen Mesh
Brief Title: Evaluate and Compare the Rate of Para-Stomal Herniation After Permanent Stoma Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Laurie Mihalik, General Surgery Clinical Study Coordinator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1712-05
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Hernia
Keywords: stoma, hernia, mesh
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): mesh reinforcement at stoma
  Interventions: Procedure: mesh reinforcement of stoma
- Arm 1 (Active Comparator): standard stoma
  Interventions: Other: no intervention

INTERVENTIONS:
Procedure: mesh reinforcement of stoma — Patients randomized to receive mesh will undergo stoma formation and will have a 8 cm x 12 cm piece of AlloDerm graft placed as a tissue reinforcement around the stoma and extending under the midline incision. The mesh will be trimmed to provide a minimum of 3cm of overlap around the stoma in all directions. The mesh will be secured with transabdominal number one Prolene (Ethicon, Inc) sutures every 4cm around the mesh. Additional fixation will be provided with Protack spiral tacks (US Surgical, Inc) every 1cm around the mesh. The midline fascia will be closed with running number one Prolene sutures. Skin will be closed in standard fashion.
  Arms: 2
Other: no intervention
  Arms: Arm 1

SUMMARY:
This study is being done to evaluate the use of a material (Alloderm collagen mesh) during the stomal formation operation (surgery that will create a mouth-like opening on the surface of the body to an internal organ). The main purpose of this research study is to see if using this material will lower the hernia rate compared to normal repair without this material. The secondary purpose is to evaluate if using this material will increase or decrease complication rates.

DETAILED DESCRIPTION:
This study seeks to examine the ability of an implantable collagen matrix to reduce the incidence of parastomal hernia formation. Patients will be randomized preoperatively by a computer generated random allocation to either receive collagen mesh at the time of stoma formation, or to have stoma formation without mesh. Stomas without mesh will be made in the standard surgical fashion dictated by the type of stoma: ileostomy, colostomy, ileal conduit. Patients randomized to receive mesh will undergo stoma formation in an identical fashion, and will have a 8 cm x 12cm piece of AlloDerm mesh placed as a tissue reinforcement at the stoma site and extending under the midline incision. Patients will be followed with physical examinations at approximately 2weeks post-op, 3, 6, 9, 12, 24 months post-op, and will undergo CT scanning of the abdomen and pelvis at 12 and 24months to determine hernia occurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be at least 18 years of age.
2. Male or female (excluding pregnant females).
3. Patients will require stoma formation.
4. Patients with ASA < 3.
5. Patients informed about the study, and will have read; understood and signed the patient informed consent and authorization to use their PHI, as applicable.
6. Patients will be willing and able to submit to postoperative follow-up evaluations.

Exclusion Criteria:

1. Patients that have had prior surgical treatment parastomal herniation.
2. Patients that refuse stoma formation.
3. Patients with ASA > 3.
4. Patients who have certain metabolic conditions (e.g., chronic hepatic or renal disease).
5. Patients with evidence of pre-existing systemic or local infections.
6. Patients with wound-healing or autoimmune disorders.
7. Patients who, in the surgeon's opinion, would have a difficult time comprehending or complying with the requirements of the study.
8. Patients with any conditions that were not suspected preoperatively and are only discovered at the time of the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Rate of parastomal hernia formation. | 2 years post-op

CONTACTS AND LOCATIONS:
Overall Officials: Kristi L Harold, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States